CLINICAL TRIAL: NCT00611988
Title: Self-Managed Walking Improves Function in Patients With Diabetes Mellitus and Peripheral Arterial Disease
Brief Title: Self-Managed Walking Improves Function
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Kansas (Other)
Collaborators: American Diabetes Association (Other)
Responsible Party: Principal Investigator, Tracie Collins, MD, MPH, Prinicpal investigator, University of Kansas
Organization: University of Kansas Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 0607M89406; 7-06-CR-10
Record Dates: First submitted 2008-01-25; First posted 2008-02-11 (Estimated); Last update posted 2013-12-10 (Estimated); Status verified 2013-12

CONDITIONS: Peripheral Arterial Disease; Diabetes Mellitus
Keywords: Walking therapy; Diabetes mellitus; Peripheral arterial disease
MeSH Terms: conditions — Peripheral Arterial Disease; Diabetes Mellitus | interventions — Control Groups

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): The intervention includes individual therapy, group reinforcement, and follow-up phone contact
  Interventions: Behavioral: Self-managed walking
- 2 (Active Comparator): Attention control group will receive routine follow-up phone calls
  Interventions: Other: Control group

INTERVENTIONS:
Behavioral: Self-managed walking — The intervention includes individual therapy, group reinforcement, and follow-up phone contact
  Other Names: behavorial intervention
  Arms: 1
Other: Control group — Attention control group will receive routine follow-up phone calls
  Other Names: Attention control
  Arms: 2

SUMMARY:
We are conducting a clinical research trial to determine the role of self-managed walking therapy to improve walking ability in patients with diabetes mellitus and peripheral arterial disease (PAD). PAD, commonly referred to as poor circulation in the legs, is a very common disease in patients with diabetes mellitus. For patients with PAD, there is a significant risk for poor walking ability and limb loss. One major treatment for PAD is walking therapy but the traditional methods for the delivery of this treatment have required frequent visits to a university or hospital-based site. We will address the role of self-managed walking program, to be conducted at or near the home, to improve limb function.

DETAILED DESCRIPTION:
Peripheral arterial disease (PAD) is a prevalent illness that affects 12% of U.S adults. Diabetes mellitus is one of the strongest atherosclerotic risk factors for this disease. Among patients with diabetes mellitus, the prevalence of PAD is as high as 29%. An underutilized component of care for PAD is walking therapy. Walking has specifically been shown to improve functional status in patients with PAD and leg symptoms.

Leg symptoms in PAD include intermittent claudication and atypical leg symptoms (leg discomfort other than intermittent claudication). Patients with symptomatic PAD have impaired lower extremity functioning, which clinically manifests as slower walking speed, reduced walking distance, and lower physical activity levels. These functional deficits often hinder the ability to live independently in the community (e.g., walking to the bus stop in time for the next bus, shopping independently for groceries). Reduced physical activity is associated with an increased risk for mobility loss and a higher risk for functional decline with subsequent inability to perform activities of daily living.

Walking therapy should not be a burden and it should be something that the patient can routinely perform without the need for regular supervision, a treadmill, or to report to the hospital (i.e., self-managed walking therapy). As patients with diabetes mellitus have special needs for self-management behavior (e.g., diet, medication adherence) and, for those with PAD, a higher burden of atypical leg symptoms, the role of a self-managed walking program specific to this group of PAD patients cannot be overemphasized. Thus, this clinical trial has 2 novel aspects: 1) to evaluate the role of self-managed walking therapy for patients with symptomatic PAD and 2) to focus on patients with PAD and diabetes mellitus.

ELIGIBILITY:
Inclusion Criteria:

* Age 40 years and older
* Diabetes mellitus
* Peripheral arterial disease
* Leg symptoms

Exclusion Criteria:

* Myocardial infarction within 3 months of enrollment
* Inability to walk for exercise secondary to chest pain, dyspnea, or poor balance
* Prior major amputation

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 145 (Actual)
Dates: Start 2006-08; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
Maximal treadmill walking distance | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Tracie C Collins, MD, Principal Investigator — University of Kansas Medical Center
Locations (1):
- KU School of Medicine - Wichita, Wichita, Kansas, United States

REFERENCES:
- [Derived] Collins TC, Lunos S, Carlson T, Henderson K, Lightbourne M, Nelson B, Hodges JS. Effects of a home-based walking intervention on mobility and quality of life in people with diabetes and peripheral arterial disease: a randomized controlled trial. Diabetes Care. 2011 Oct;34(10):2174-9. doi: 10.2337/dc10-2399. Epub 2011 Aug 26. PMID 21873560